CLINICAL TRIAL: NCT01441271
Title: Diverting Loop Ileostomy and Colonic Lavage: An Alternative To Total Abdominal Colectomy For The Treatment Of Fulminant Clostridium Difficile Colitis. A Randomized Controlled Trial.
Brief Title: Optimal Surgical Treatment Of Fulminant Clostridium Difficile Colitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Numer of eligible patients markedly decreased since the initiation of the study.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Marc A. de Moya, Assistant Professor of Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-P-000138/1; MGH
Record Dates: First submitted 2011-09-17; First posted 2011-09-27 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Clostridium Difficile Colitis
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — Therapeutic Irrigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- total abdominal colectomy (Active Comparator): the standard of care for fulminant clostridium difficile colitis is a total abdominal colectomy
  Interventions: Procedure: total abdominal colectomy
- Ileal diversion and lavage (Experimental): The tested intervention in this trial will be: intraoperative colonic lavage using a high volume polyethylene glycol/electrolyte solution, that will clear Clostridium difficile infection resulting in eradication of FCDC while preserving the colon.
  Interventions: Procedure: Ileal diversion and lavage

INTERVENTIONS:
Procedure: Ileal diversion and lavage — The surgical approach involves an attempted laparoscopic creation of a loop ileostomy after visually assessing the colon to assure viability. If the loop is unable to be safely performed laparoscopically an open loop ileostomy will be performed. Intraoperatively, 8 liters of warmed polyethylene glycol 3350/electrolyte solution [GoLytely®; Braintree Laboratories] will be infused into the colon via the ileostomy and collected via a rectal drainage tube. Post-operatively, the patients will receive antegrade vancomycin flushes [500 mg in 500 ml of Lactated Ringers; q8 hours for duration of 10 days] via a Malecot catheter [24 French] left in the efferent limb of the ileostomy (Figure 1). Additionally patients will be continued on intravenous metronidazole [500mg q8 hours] for 10 days.
  Arms: Ileal diversion and lavage
Procedure: total abdominal colectomy — The surgical approach of the colon in a total abdominal colectomy involves a midline incision. The complete colon in the abdomen (from ileum to rectum) will be removed and an end ileostomy is performed.
  Other Names: subtotal colectomy
  Arms: total abdominal colectomy

SUMMARY:
The investigators hypothesize that minimally invasive ileal diversion with intraoperative colonic lavage using a high volume polyethylene glycol/electrolyte solution will clear Clostridium difficile infection resulting in eradication of Fulminant C. difficile colitis (FCDC) while preserving the colon. Furthermore, the investigators hypothesize this will reduce morbidity and mortality compared to total abdominal colectomy.

DETAILED DESCRIPTION:
Clostridium difficile (C. difficile) affects more than 3 million patients per year in the United States, and is increasing in frequency [2-15]. Approximately 8 % of hospitalized patients are infected with C. difficile [12]. Of these patients 3% - 8% will develop the fulminant disease, defined as C. difficile colitis with significant systemic toxic effects and shock, resulting in need for colectomy or death [2].

Fulminant C. difficile colitis (FCDC) is a highly lethal disease with mortality rates ranging between 12% - 80% [2-6,8-15]. A retrospective study in our own institution identified a 35% mortality rate for FCDC [2].

The indications for surgical management of patients with FCDC are not clearly defined, however most advocate surgical intervention in patients with worsening clinical exams, peritonitis, or patients in shock. Total abdominal colectomy (also called subtotal colectomy) with end ileostomy has been advocated as the operation of choice and has been demonstrated to marginally improve survival compared to non-operative management in these critically ill patients. A total abdominal colectomy has many disadvantages. Most important, mortality rates continue to range from 35-80%. Additionally, total abdominal colectomy (subtotal colectomy) can result in significant morbidity, and many survivors will have a permanent ileostomy.

The new treatment option that will be tested in this randomized controlled trial (RCT) may change the standard of care. Based on a small prospective series from Neal and colleagues [1] the investigators propose an alternative surgical approach for the management of FCDC, which may prove a safer and simpler option. Based on the nature of the disease as a bacterial toxin-mediated mucosal inflammatory process with delayed and indirect systemic threats to life, the investigators think that minimally invasive ileal diversion with intraoperative colonic lavage using a high volume polyethylene glycol/electrolyte solution will clear Clostridium difficile infection resulting in eradication of FCDC while preserving the colon.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients >18 years of age
2. Able to provide informed consent, or presence of a legally authorized representative able and willing to provide informed consent
3. Candidates for total abdominal colectomy due to severe, complicated FCDC per consulting surgeon and team providing care
4. Subjects must meet criteria for operative management of FCDC (find in detailed protocol)

Exclusion Criteria:

1. Children (<18 years of age)
2. Allergy or hypersensitivity reaction to study medications: Vancomycin, Metronidazole, GoLytely
3. Intra-operative evidence of colonic perforation
4. Intra-operative evidence of colonic necrosis
5. Pregnancy (this will be ruled out by a urine test at the time of indication for surgery)
6. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 day
  Both groups will be compared using mortality as the primary outcome.

SECONDARY OUTCOMES:
ICU Length of Stay (LOS | during hospitalization
  14 days
Hospital LOS | hospitalization
  1 year
ventilation days | while in ICU
  1 year
morbidity | during hospitalization
  1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marc de Moya, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States